CLINICAL TRIAL: NCT01819220
Title: Randomized, Open Labeled Clinical Trial to Compare the Effectiveness of Amlodipine/Valsartan vs Hydrochlorothiazide/Telmisartan on Glucose Tolerance in Patients With Hypertension With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2009-0077
Record Dates: First submitted 2013-03-15; First posted 2013-03-27 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination; Valsartan; telmisartan, hydrochlorothiazide drug combination; Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- amlodipine/valsartan (Active Comparator)
  Interventions: Drug: amlodipine/valsartan
- hydrochlorothiazide/telmisartan (Experimental)
  Interventions: Drug: hydrochlorothiazide/telmisartan

INTERVENTIONS:
Drug: amlodipine/valsartan — This is a phase IV clinical study. The study is a 24 week, prospective, randomized open labeled multicenter study to compare the efficacy of amlodipine/valsartan combination vs telmisartan/hydrochlorothiazide combination in reducing post prandial sugar. The study will be performed in hypertensive patients with metabolic syndrome.
  Active group: Starting dose of amlodipine 5mg/ valsartan 80mg comparator group: Telmisartan 40mg/hydrochlorothiazide 12.5mg When the blood pressure is above the target goal of 140/90mmHg, up titration to amlodipine 5/valsartan 160 and/or telmisartan 80/hydrochlorothiazide 12.5mg is allowed.
  When the blood pressure is above 140/90mmhg at the 12th week, addition of doxazosin 4mg is allowed.
  Other Names: Starting dose of amlodipine 5mg/ valsartan 80mg
  Arms: amlodipine/valsartan
Drug: hydrochlorothiazide/telmisartan — When the blood pressure is above the target goal of 140/90mmHg, uptitration to amlodipine 5/valsartan 160 and/or telmisartan 80/hydrochlorothiazide 12.5mg is allowed.
  When the blood pressure is above 140/90mmhg at the 12th week, addition of doxazosin 4mg is allowed.
  Other Names: Telmisartan 40mg/hydrochlorothiazide 12.5mg
  Arms: hydrochlorothiazide/telmisartan

SUMMARY:
Recent studies have demonstrated that RAS inhibitors/calcium channel blockers are superior to RAS inhibitors/diuretics for reducing cardiovascular outcomes in hypertension. As such, RAS inhibitors/calcium channel blockers are recommended as first line combination treatment for hypertension. However, the mechanism for the superior efficacy of RAS inhibitors/calcium channel blockers are not well defined. This study will compare the efficacy of RAS inhibitors/calcium channel blockers vs RAS inhibitors/diuretics in terms of glucose tolerance and insulin resistance in hypertensive patients with metabolic syndrome. The primary endpoint will be that RAS inhibitors/calcium channel blockers will be more efficacious in reducing 2hour post prandial glucose compared to RAS inhibitors/diuretics.

ELIGIBILITY:
Inclusion Criteria:

* consent to the study
* Male or Female ≥ 20 years
* Patients taking less than 1 antihypertensive medications or not taking antihypertensive medications. Hypertension defined at the screening visit as follows): 140mmHg < MSSBP or MSDBP > 90mmHg at screening
* Hypertensive patients with non diabetic metabolic syndrome will be enrolled. Metabolic syndrome is defined according to NCEP guideline. (3 or more than) ① Abdominal obesity: Waist circumference M ≥ 90cm, F ≥ 80cm

  ② Hypertriglyceridaemia: Triglycerides ≥ 150mg/dL

  ③ Low HDL cholesterol Men: HDL cholesterol ≤ 40mg/dL Women: HDL cholesterol ≤ 50mg/dL

  ④ Elevated blood pressure (systolic blood pressure ≥ 130 mmHg and diastolic blood pressure ≥ 85 mmHg, or current use of antihypertensive drugs)

  ⑤ Impaired fasting glucose: fasting plasma glucose ≥ 100 mg/dL
* Patient not taking statin medication and if the patient had ate statin medication the last duration must be before 3 months.

Exclusion Criteria:

* • Women of child-bearing potential without a contraceptive measure

  * (Pregnant or nursing women
  * Known or suspected contraindications: history of allergy or hypersensitivity
  * History of clinically significant allergies including asthma and/or multiple drug allergies
  * Patients taking more than 2 antihypertensive medications
  * Patient taking statin medication and taking statin within 3 months
  * MSSBP > 180 mmHg or MSDBP > 110 mmHg at any time during the study
  * Evidence of a secondary form of hypertension)
  * History of hypertensive encephalopathy, cerebrovascular accident, transient ischemic attack, myocardial infarction, percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG) for 12 months prior to Visit 1
  * History of heart failure Grade II - IV according to the NYHA classification
  * Concomitant potentially life threatening arrhythmia or symptomatic arrhythmia
  * Concomitant unstable angina pectoris
  * Clinically significant valvular heart disease
  * Patients with Type 1 or Type 2 diabetes mellitus
  * Evidence of hepatic disease as determined by one of the following: AST or ALT values ≥ 3 x UNL, a history of hepatic encephalopathy, history of esophageal varices, or history of portocaval shunt
  * Evidence of renal impairment as determined by one of the following: serum creatinine >2mg/dL , history of dialysis, or history of nephrotic syndrome
  * Protein in U/A values 2+ ≤
  * Serum potassium values < 3.2 or > 5.2 mmol/L
  * History of malignancy of any organ system within the past 5 years, treated or untreated, including leukemia and lymphoma, as further defined in the full protocol
  * Chronic use of NSAIDs
  * Use of cyclooxygenase-2 inhibitors (COX-2 inhibitors
  * Use of niacin > 100 mg/d
  * Use of loop diuretics
  * Use of statin shorter than 3 months
  * Inability to discontinue prior antihypertensive drugs as specified in the full protocol
  * persons directly involved in the execution of this protocol
  * Volume depletion based on the investigator's clinical judgment using vital signs, skin turgor, moistness of mucous membranes, and laboratory values
  * Any severe, life-threatening disease within the past five years

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To assess the glucose change | To assess the change from baseline (week 0) to study endpoint (week 24) on 2hr-post-prandial plasma glucose level using oral glucose tolerance test (75-g OGTT)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei universty medical center, Seoul, Seoul, South Korea